CLINICAL TRIAL: NCT04145375
Title: Continuation Protocol for ZEN003694 in Patients Experiencing Clinical Benefit While Enrolled in a ZEN003694 Protocol
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zenith Epigenetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEN003694-500
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: mCRPC
Keywords: Zenith; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: ZEN003694 in Combination with Enzalutamide (Experimental): Patients who have completed participation in their original ZEN003694-002 protocol and have clinical benefit as determined by the investigator may continue to receive treatment with ZEN003694 in combination with enzalutamide
  Interventions: Drug: ZEN003694; Drug: Enzalutamide

INTERVENTIONS:
Drug: ZEN003694 — Up to 120mg
Drug: Enzalutamide — 160mg
  Other Names: Xtandi; MDV3100

SUMMARY:
Continuation Protocol for ZEN003694 in Patients Experiencing Clinical Benefit While Enrolled in a ZEN003694 Protocol

DETAILED DESCRIPTION:
This is an open label, non-randomized, single-arm continuation protocol study using ZEN003694. Patients who have completed participation in their original ("parent") ZEN003694 protocol and have clinical benefit as determined by the investigator may continue to receive treatment with ZEN003694 in the continuation protocol. The patient must have been enrolled in a Zenith Epigenetics sponsored ZEN003694 therapeutic study to be eligible for participation in this continuation protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Protocol-defined completion in a parent ZEN003694 trial
2. Patient has clinical benefit as determined by the investigator at the time of entry to the continuation protocol
3. ECOG performance status of 0 or 1
4. Acceptable ZEN003694 tolerability, in the judgment of the investigator
5. Initiation of dosing in this continuation trial to occur within two weeks (14 days) of completing dosing in the parent trial, unless more time is approved by the sponsor in writing

Exclusion Criteria:

1. Concurrent participation in another clinical investigational treatment trial
2. Require addition of or change to a new concomitant therapy to adequately treat the malignancy under study
3. Discontinued ZEN003694 or withdrew consent to participate in original Zenith Epigenetics-sponsored ZEN003694 study
4. Any other reason that in the opinion of the Investigator would prevent the patient from completing participation or following the study schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events (AE) and treatment-related serious adverse events (SAE) | Up to 3 years

SECONDARY OUTCOMES:
Evaluate radiographic response rate by RECIST 1.1 criteria | Up to 3 years
Evaluate Overall survival (OS): Time from date of first dose of ZEN003694 in the parent protocol or randomization to the date of death from any cause | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California San Francisco Medical Center, San Francisco, California
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No